CLINICAL TRIAL: NCT00001280
Title: Itraconazole for the Prevention of Fungal Infections in Chronic Granulomatous Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 910064; 91-I-0064
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Mycoses
Keywords: Aspergillosis; Phagocyte Defect; Torulopsis; Chronic Granulomatous Disease
MeSH Terms: conditions — Mycoses; Aspergillosis; Torulopsis; Granulomatous Disease, Chronic | interventions — Itraconazole

INTERVENTIONS:
Drug: itraconazole

SUMMARY:
This protocol describes a prospective, randomized study examining the safety and efficacy of Itraconazole for preventing fungal infections in patients with Chronic Granulomatous Disease (CGD). CGD is a genetic disorder in which phagocytes are unable to produce oxygen radicals. As a result, affected patients are prone to recurrent, severe infections with bacterial and fungal organisms. Patients with CGD of 5 or more years of age without evidence of infection at the time of study entry will be eligible for enrollment. Patients will be randomized to receive itraconazole or placebo tablets daily, in a double blinded fashion. In addition to itraconazole, all patients will receive antimicrobial prophylaxis against bacterial infection, and may in addition receive gamma-interferon as prophylaxis against infection. Randomization of patients will be stratified among patients receiving or not receiving gamma interferon. The primary endpoint of the study will be the development of culture or histologically proved invasive fungal disease. Patients will be monitored every three months for evidence of drug toxicity. The anticipated accrual period will be approximately 36-48 months.

DETAILED DESCRIPTION:
This protocol describes a prospective, randomized study examining the safety and efficacy of Itraconazole for preventing fungal infections in patients with Chronic Granulomatous Disease (CGD). CGD is a genetic disorder in which phagocytes are unable to produce oxygen radicals. As a result, affected patients are prone to recurrent, severe infections with bacterial and fungal organisms. Patients with CGD of 5 or more years of age without evidence of infection at the time of study entry will be eligible for enrollment. Patients will be randomized to receive itraconazole or placebo tablets daily, in a double blinded fashion. In addition to itraconazole, all patients will receive antimicrobial prophylaxis against bacterial infection, and may in addition receive gamma-interferon as prophylaxis against infection. Randomization of patients will be stratified among patients receiving or not receiving gamma interferon. The primary endpoint of the study will be the development of culture or histologically proved invasive fungal disease. Patients will be monitored every three months for evidence of drug toxicity, and surveillance cultures of nasopharynx and stool will be obtained. The anticipated accrual period will be approximately 36-48 months.

ELIGIBILITY:
Documented chronic granulomatous disease more than 5 years of age.

No fungal infection within the past year.

Not currently on other antifungals or have taken other antifungals during the past 3 months.

Not currently on phenytoin or rifampin.

Negative pregnancy test within 2 weeks of starting protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1991-01; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hardin TC, Graybill JR, Fetchick R, Woestenborghs R, Rinaldi MG, Kuhn JG. Pharmacokinetics of itraconazole following oral administration to normal volunteers. Antimicrob Agents Chemother. 1988 Sep;32(9):1310-3. doi: 10.1128/AAC.32.9.1310. PMID 2848442
- [Background] Gallin JI, Buescher ES, Seligmann BE, Nath J, Gaither T, Katz P. NIH conference. Recent advances in chronic granulomatous disease. Ann Intern Med. 1983 Nov;99(5):657-74. doi: 10.7326/0003-4819-99-5-657. PMID 6227266